CLINICAL TRIAL: NCT04001816
Title: A Randomized Clinical Trial to Investigate Whether Self Ligating Brackets or Conventional Brackets Are Better for Treating Bimaxillary Proclination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Collaborators: University of Dundee (Other)
Responsible Party: Principal Investigator, Trudee Hoyte, Principal Investigator, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UWestIndiesSt.Augustine
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Bimaxillary Proclination
MeSH Terms: interventions — Orthodontic Brackets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Orthodontic Brackets — Self ligating and Conventional brackets

SUMMARY:
The study is a single blind randomised control trial.The patients will be randomly assigned to have conventional brackets placed or self ligating brackets placed.

All patients will undergo full Orthodontic records. This will include an Orthodontic assesment, study models relevant xrays (orthopantogram and a cephalomgram) and clinical photos. After records analysis, patients will be given a prophylaxis and oral hygiene instructions.

Either 3m Victory Series™ Metal Braces or 3m SmartClip™ SL3 Self-Ligating Braces both bracket types will carry the MBT prescription 0.022 slot height, will be bonded using Transbond™ XT (3M Unitek, Monrovia, California, USA) composite resin according to the manufactuer's instruction.

These patients will be recalled at monthly intervals for the duration of treatment time which will be 3 years. A cephalogram will be taken at the end of treatment

ELIGIBILITY:
Inclusion Criteria:

* Bimaxillary Proclination
* Class I or Class II division 1 incisor relationship with an overjet less than or equal to 6.0 mm
* The cases can be extraction or non extraction cases
* Extraction cases must be of at least both upper first premolars to relieve moderate to severe crowding and/or to reduce the overjet
* No previous orthodontic treatment
* No systemic illness
* No use of anti inflammatory drugs prior to placement of the fixed appliance
* Good oral hygiene and periodontal health with periodontal pockets of less than or equal to 4 mm, full-mouth plaque score less than or equal to 20 per cent
* Cooperative and motivated
* In the permanent dentition with all teeth present at least to the first molars
* No radiographic bone loss was observed on the dental pantomographic image.

Exclusion criteria:

* Patients who required surgery to correct skeletal discrepancies.
* Patients with hyperdontia, hypodontia, or syndromic diseases (e.g. cleft lip and palate).
* Uncooperative patients

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment time | 18-24 months
  Length of time each bracket takes to treat a bimaxillary proclination patient

CONTACTS AND LOCATIONS:
Overall Officials: Trudee Hoyte, Principal Investigator — The University of The West Indies
Locations (1):
- UWI Dental School, Saint Augustine, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: No